CLINICAL TRIAL: NCT06046131
Title: Clinical, Genetic and Environmental Determinants of Prostate Cancer Progression.
Acronym: KP-CARAIBES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PAP_RIPH2_2020/26
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Prostatic Neoplasm; Adenocarcinoma; Neoplasm Recurrence; Neoplasm Metastasis
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Recurrence; Neoplasm Metastasis | interventions — Standard of Care; Urine Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Any patient with a histologically confirmed incident case of prostate cancer will be included in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients prostate cancer (Other): Patient with a confirmed diagnosis of prostate cancer will be included before starting any treatment. Recruitment will be carried out by urologists from the urology departments of the CHU of Guadeloupe and the CHU of Rennes.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — Extra blood collection for dosages Urine collection for the dosage of non-persistent pollutants, isolation of extracellular vesicles released in urine, analysis of the microbiome, metagenomics to obtain a complete description of the bacterial functions represented as well as other microorganisms present, metabolome profiling and identification and/or assays of any other biological compound of interest strictly related to the specific objectives of the research.
  Saliva collection for the extraction of the constitutional DNA. An interview using a structured questionnaire A quality of live auto-questionnaire
  Other Names: Extra blood collection, urine collection and saliva collection, questionnaire.

SUMMARY:
The course and progression of prostate cancer is highly variable, depending on the individual characteristics, the aggressiveness of the disease at the time of diagnosis as well as the ethno-geographic origins of the individuals. The general objective of the project is to identify the clinical, genetic and environmental determinants (risk factors) of the evolution, progression and complications of the disease according to the treatment options. Identifying modifiable and non-modifiable prognostic determinants of disease progression is a major challenge. This knowledge will help guide treatment choices but also, especially in high-risk populations (high incidence of disease) to better tailor prevention policies and possibly screening .

DETAILED DESCRIPTION:
There is a lack of information to predict the course of prostate cancer following its initial diagnosis; in other words, why some are indolent and evolve very slowly and others are aggressive, evolve rapidly with an increased risk of metastasis development and death. In addition, these evolutions do not seem similar according to ethno-geographic origins. We therefore hypothesize that in addition to genetic susceptibility factors specific to individuals and / or linked to their ethno-geographic origins, medical, occupational and environmental factors can influence the course of the disease and the response to treatments. We will build two prospective cohorts of incident cases of prostate cancer, one in Guadeloupe (whose population is predominantly Afro-descendant) and one in Rennes (Brittany, whose population is mainly of Caucasian origin). Each patient will be subject to longitudinal follow-up over time. Structured questionnaires will be administered at the time of diagnosis and at regular times after the initial treatment or subsequent treatments. They will focus on socio-demographic data, places of residence, education levels, lifestyles (tobacco, alcohol), personal and family medical history, current treatments, current and past occupational activities. Anthropometric and blood pressure measurements will be made at the time of diagnosis and at regular times after treatment. Saliva, urine and blood samples will be obtained. Clinical data related to the disease will be collected continuously.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

Adult patients with incident case of prostate cancer Patient consulting the University Hospital of Guadeloupe or the University Hospital of Rennes Patient who resides in the departments of Guadeloupe or Martinique or the community of Saint-Martin or in Britany Patient affiliated or beneficiary of the social security signed consent

Exclusion Criteria:

Physical or mental health judjed by the investigator as precluding participation in the research Protected adults (guardianship, curatorship, safeguard of justice).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2039-02-28 (Estimated); Study Completion 2039-02-28 (Estimated)

PRIMARY OUTCOMES:
association between determinants (independent variables) and health events linked to disease progression (dependent variables) | At the start of the study, at 1,2,5 and 10 years after the inclusion and after starting treatment.
  dependent variables: These are mainly criteria relating to :Discharge from active surveillance, Biological recurrence,Radiological, loco-regional or distant progression,
  Independant variables. These are mainly criteria relating to :
  Date of initial treatment and dates of successive treatments, Gleason score (ISUP) at diagnosis Gleason score (ISUP) on surgical specimen pTNM stage after surgery Body mass index [kg/m²], percentage of fat mass, % of water mass, % of bone mass estimated by bio-impedance.
  Metabolic syndrome (3 of the following 5 criteria): triglycerides > 1.7 mmo

SECONDARY OUTCOMES:
association between determinants (independent variables) and health events other than those linked to disease progression (dependent variables). | : At the start of the study, at 1,2,5 and 10 years after the inlcusion and after starting treatment.
  Dependent variables Adverse events (disease-related or treatment-related) rated according to CTCAE grades (Common Terminology Criteria for Adverse Events) Micturition disorders estimated by the International Prostate Symptom Score (IPSS) Erectile function estimated by the IIEF5 score (International Index of Erectile Function) Quality of life estimated by the FACT-P score (Functional Assessment of Cancer Therapy-Prostate) Independent variables These are the same as those indicated for the primary endpoints.

CONTACTS AND LOCATIONS:
Locations (2):
- CHU of Rennes, Rennes, Ille-et-Vilaine, France
- CHU of Guadeloupe, Pointe-à-Pitre, Guadeloupe, Guadeloupe